CLINICAL TRIAL: NCT00908349
Title: Multicenter, Open-Label Extension Study to Evaluate the Long-Term Safety and Tolerability of OXC XR as Adjunctive Therapy in Subjects With Refractory Partial Epilepsy
Brief Title: Safety and Tolerability of OXC XR as Adjunctive Therapy in Subjects With Refractory Partial Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 804P302
Record Dates: First submitted 2009-05-22; First posted 2009-05-25 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Partial Epilepsy
MeSH Terms: conditions — Epilepsies, Partial | interventions — Oxcarbazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxcarbazepine XR (Other): Open Label Study
  Interventions: Drug: Oxcarbazepine XR

INTERVENTIONS:
Drug: Oxcarbazepine XR — Open Label Study
  Other Names: SPN-804O

SUMMARY:
Open-Label Extension Study to Evaluate the Long-Term Safety and Tolerability of Oxcarbazepine Extended-Release (OXC XR)

DETAILED DESCRIPTION:
NAP

ELIGIBILITY:
Inclusion Criteria

1. Able to provide written informed consent and agree to comply with study procedures.
2. Male or female aged 18 to 66 years, inclusive.
3. Successful completion of the 804P301 study.
4. Sexually active women, unless surgically sterile (at least 6 months prior to Study Medication [SM] administration) or at least 1 year post-menopausal, must use an effective method of avoiding pregnancy (including oral, transdermal, or implanted contraceptives [any hormonal method in conjunction with a secondary method], intrauterine device, female condom with spermicide, diaphragm with spermicide, cervical cap, abstinence, use of condom with spermicide by sexual partner or sterile [at least 6 months prior to SM administration] sexual partner) for at least four weeks prior to SM administration, and must agree to continue using such precautions through the End of Study visit. Cessation of birth control after this point should be discussed with a responsible physician.

Exclusion Criteria

1. Clinically significant change in health status that, in the opinion of the Investigator, would prevent the subject from participating in this study or successfully completing this study.
2. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2009-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet K Johnson, PhD, Study Director — Supernus Pharmaceuticals, Inc.
Locations (58):
- United States (20):
  - Huntsville, Alabama
  - Northport, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Riverside, California
  - West Los Angeles, California
  - Aurora, Colorado
  - Jacksonville, Florida
  - Miami, Florida
  - Sarasota, Florida
  - Springfield, Illinois
  - Lexington, Kentucky
  - Bethesda, Maryland
  - Missoula, Montana
  - New York, New York
  - Oklahoma City, Oklahoma
  - Nashville, Tennessee
  - Baytown, Texas
  - Temple, Texas
- Bulgaria (5):
  - Blagoevgrad
  - Pleven
  - Rousse
  - Sofia
  - Varna
- Canada (2):
  - Calgary, Alberta
  - Greenfield Park, Quebec
- Croatia (2):
  - Dubrovnik
  - Zagreb
- Mexico (8):
  - Col. Las Palmas, Chihuahua
  - Col. Guillermina, Durango
  - Guadalajara, Jalisco
  - Zapopan, Jalisco
  - Mexico City, Mexico City
  - San Luis Potosí City, San Luis Potosí
  - Aguascalientes
  - Puebla City
- Poland (7):
  - Giżycko
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Warsaw
  - Wilkowice
- Romania (4):
  - Bucharest
  - Campulung Muscel
  - Cluj-Napoca
  - Craiova
- Russia (10):
  - Kazan'
  - Kirov
  - Kursk
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Pyatigorsk
  - Saint Petersburg
  - Samara
  - Smolensk

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxcarbazepine XR: Oxcarbazepine XR: Open Label Study 600mg to 2400mg of SPN-804O once daily.
Period: Overall Study
Arm/Group | Oxcarbazepine XR
Started | 214
Completed | 179
Not Completed | 35
Not completed — Adverse Event | 10
Not completed — Withdrawal by Subject | 9
Not completed — Physician Decision | 5
Not completed — Lost to Follow-up | 5
Not completed — Various | 6

BASELINE CHARACTERISTICS:
Arm/Group | Oxcarbazepine XR
Number analyzed (Participants) | 214
Age, Continuous [Mean (Full Range); unit: Years] | 37.4 [18 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111
  Male | 103
Region of Enrollment [Number; unit: participants]
  United States | 43
  Mexico | 30
  Canada | 2
  Poland | 31
  Romania | 12
  Croatia | 6
  Russian Federation | 64
  Bulgaria | 26

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Seizure Rate
Description: Measured as change from baseline to end of study
Time Frame: one year
Measure: Median (Full Range); unit: percentage of change in seizure rate
Arm/Group | Oxcarbazepine XR
Number analyzed (Participants) | 214
percentage of change in seizure rate | -26.3 [-100.0 to 344.7]

ADVERSE EVENTS:
Arm/Group | Oxcarbazepine XR
Serious Adverse Events (participants affected / at risk) | 18/214
Other Adverse Events (participants affected / at risk) | 124/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxcarbazepine XR (N=214)
Hypothermia (General disorders) | 1 (1)
Spinal Fracture (Injury, poisoning and procedural complications) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Prostatic Specific Antigen Increased (Investigations) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Grand Mal Convulsion (Nervous system disorders) | 2 (2)
Non-Cardiac Chest Pain (General disorders) | 2 (2)
Epilepsy (Nervous system disorders) | 2 (2)
Suicidal Behaviour (Psychiatric disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Pyelonephritis Acute (Infections and infestations) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oxcarbazepine XR (N=214)
Dizziness (Nervous system disorders) | 33
Headache (Nervous system disorders) | 24
Diplopia (Eye disorders) | 20
Nausea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 13
Somnolence (Nervous system disorders) | 12
Balance Disorder (Nervous system disorders) | 10
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other